CLINICAL TRIAL: NCT05565664
Title: Ketamine Hydrochloride Versus Magnesium Sulfate as Analgesic Adjuvants in Pediatric Adenotonsillectomy, a Randomized Comparative Study
Brief Title: Ketamine Versus Magnesium as Analgesic Adjuvants in Pediatric Adenotonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MD-60-2022
Record Dates: First submitted 2022-09-24; First posted 2022-10-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Post Operative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Active Comparator): After preoperative assessment, participants will receive IM midazolam (0.1 mg/kg) and atropine (0.02 mg/kg) 30 min. before surgery as premedication.
  Inhalation induction of GA will be done using 8% sevoflurane in 100% oxygen. After insertion of a peripheral IV cannula, IV fentanyl 1 mcg/kg and atracurium 0.5 mg/kg will be given. Direct laryngoscopy will be attempted to insert an age-appropriate cuffed ETT.
  Patients will be maintained on controlled mechanical ventilation with a mixture of isoflurane in 60% oxygen in air, using a tidal volume of 8cc/kg and a frequency of 16-20 cycle/min. to maintain an ETCO2 35-40 mmHg and to keep an ET isoflurane concentration of 1.5-2%. All patients will receive 10 ml/kg of IV Ringer's solution in the operating room. A single dose of paracetamol 15 mg/kg IV drip will be administered for all patients once they arrive at the PACU.
  Patients will receive IV ketamine hydrochloride in a dose of 0.5 mg/kg.
  Interventions: Drug: Ketamine hydrochloride
- Magnesium group (Active Comparator): After preoperative assessment, participants will receive IM midazolam (0.1 mg/kg) and atropine (0.02 mg/kg) 30 min. before surgery as premedication.
  Inhalation induction of GA will be done using 8% sevoflurane in 100% oxygen. After insertion of a peripheral IV cannula, IV fentanyl 1 mcg/kg and atracurium 0.5 mg/kg will be given. Direct laryngoscopy will be attempted to insert an age-appropriate cuffed ETT.
  Patients will be maintained on controlled mechanical ventilation with a mixture of isoflurane in 60% oxygen in air, using a tidal volume of 8cc/kg and a frequency of 16-20 cycle/min. to maintain an ETCO2 35-40 mmHg and to keep an ET isoflurane concentration of 1.5-2%. All patients will receive 10 ml/kg of IV Ringer's solution in the operating room. A single dose of paracetamol 15 mg/kg IV drip will be administered for all patients once they arrive at the PACU.
  Patients will receive IV magnesium sulphate in a dose of 40 mg/kg.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Ketamine hydrochloride — Ketamine hydrochloride will be made in a 20 ml syringe in a concentration of 1.25 mg/ml. Patients will receive IV ketamine hydrochloride in a dose of 0.5 mg/kg (equivalent to 0.4 ml/kg) over 10 min.
  The coordinator of the study will prepare blinded syringes for each group, while the anesthetist who will be in charge of anesthetic management during the operation will be unaware of the study medication.
  Arms: Ketamine group
Drug: Magnesium sulfate — A 20 ml syringe will contain magnesium sulphate in a concentration 100 mg/ml (10%). Patients will receive 40 mg/kg of IV magnesium sulphate (equivalent to 0.4 ml/kg) over 10 min.
  The coordinator of the study will prepare blinded syringes for each group, while the anesthetist who will be in charge of anesthetic management during the operation will be unaware of the study medication.
  Arms: Magnesium group

SUMMARY:
Adeno-tonsillectomy is one of the most common surgeries in children. The most common complication associated is postoperative pain. If not well controlled, especially in preschool children, it can lead to a longer recovery period, delayed discharge, and nutritional deficiencies resulting in dehydration. These factors will increase hospitalization period and the need for intravenous fluids.

For this purpose, a large number of studies has been designed to evaluate the analgesic effects of various drugs during the perioperative period. Opioids are associated with sedation and respiratory depression, NSAIDs increase the risk of reoperation for bleeding while local anesthetics may cause vasoconstriction of the operation site.

For several years, N-methyl-D-aspartate (NMDA) receptors antagonists, such as ketamine and magnesium, have been used successfully to decrease postoperative pain and analgesic requirements in adult patients undergoing a number of different procedures. Ketamine reduces the needed analgesia after tonsillectomy. Most studies have shown that ketamine administration has no side effects such as hemodynamic, respiratory complications and airway problems.

Magnesium is a physiological antagonist of the NMDA receptor ion channel that plays a key role in central sensitization. Many studies have investigated the effect of magnesium sulphate on postoperative pain and opioid consumption. However, results of those studies were variable. Whereas most studies describe the reduction of postoperative analgesic requirements after magnesium sulfate, a few studies show insignificant beneficial effects.

A previous study evaluated the effect of low dose ketamine (0.15 mg/kg) and magnesium sulfate (30 mg/kg) on post tonsillectomy pain in children, which did not demonstrate a decrease in pain or analgesic consumption in children undergoing tonsillectomy. In this study, the investigators will increase the dose of ketamine to (0.5 mg/kg) and magnesium sulfate to (40 mg/kg) to evaluate their effect on postoperative pain in pediatric patients undergoing adeno-tonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders.
2. American society of anesthesiologists (ASA) physical status class I and ll.
3. Patients undergoing adeno-tonsillectomy.

Exclusion Criteria:

1. Inability to provide an informed consent.
2. Patients with suspected difficult airway.
3. History of allergy to ketamine or magnesium.
4. Metabolic and endocrine disorders.
5. Growth developmental, and motor-mental retardation.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
The postoperative pain score | 6 hours after surgery
  The postoperative pain score after adeno-tonsillectomy using modified Children's Hospital Eastern Ontario Pain Scale (CHEOPS). It is a behavioral scale that includes 6 categories (each has a score from 0 to 2): cry, facial, verbal, torso, legs and touch (with a total score range from 0 to 12). Higher scores mean worse outcome (higher pain intensity).

SECONDARY OUTCOMES:
Extubation time | time from discontinuation of volatile anesthetic agent till patient extubation when fully awake, 30 minutes after end of surgery
  The duration between the end of anesthesia and extubation
Recovery time | 1 hour after end of surgery
  the period in minutes from extubation until patient reaches a score of 9 or higher according to modified Aldrete score, when the patients will be ready to transfer to the ward
Heart rate | before induction of anesthesia, 1 minute before intubation, 1 minute after intubation, every 10 min intraoperatively, 1 minute before extubation, at admission to post-anesthesia care unit (PACU), 15 and 30 min after PACU admission
  Preoperative, intraoperative and postoperative heart rate (beats per minute)
Mean arterial blood pressure | before induction of anesthesia, 1 minute before intubation, 1 minute after intubation, every 10 min intraoperatively, 1 minute before extubation, at admission to post-anesthesia care unit (PACU), 15 and 30 min after PACU admission
  Preoperative, intraoperative and postoperative mean arterial blood pressure (in mmHg)
Postoperative nausea and vomiting in the PACU | 1 hour after end of surgery
  The incidence of postoperative nausea and vomiting in the PACU (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Jehan Elkholy, M.D., Study Chair — Cairo University; Eman Fouad Ali, M.D., Study Director — Cairo University; Kareem MA Nawwar, M.D., Study Director — Cairo University; Mohamed A Ashour, M.Sc., Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt